CLINICAL TRIAL: NCT01066793
Title: Prospective Observational Study on Predictors of Early On-treatment Response and Sustained Virological Response in a Cohort of Treatment naïve HCV-infected Patients Treated With Pegylated Interferons.
Brief Title: PROPHESYS 2: An Observational Study on Predictors of Response in Treatment-naïve Patients With Chronic Hepatitis C Treated With Pegasys (Peginterferon Alfa-2a) or Peginterferon-alfa-2b
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MV21020
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Participants chronically infected with the hepatitis C virus including genotypes 1 to 6
  Interventions: Drug: Peginterferon alfa-2a [Pegasys]; Drug: Peginterferon alfa-2b [PegIntron®]

INTERVENTIONS:
Drug: Peginterferon alfa-2a [Pegasys] — Peginterferon/ribavirin treatment period as prescribed by treating physician (e.g. 24 or 48 weeks) and treatment-free follow-up period of 24 weeks.
Drug: Peginterferon alfa-2b [PegIntron®] — Peginterferon/ribavirin treatment period as prescribed by treating physician (e.g. 24 or 48 weeks) and treatment-free follow-up period of 24 weeks.

SUMMARY:
This observational study will assess predictors of early on-treatment and sustained virological response in treatment-naïve patients with chronic hepatitis C initiated on treatment with Pegasys (peginterferon alfa-2a) or peginterferon alfa-2b and ribavirin. Data will be collected during the treatment period (24 or 48 weeks) and 12 and 24 weeks after the end of treatment. Target sample size is <2000.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* chronic hepatitis C
* informed consent to data collection

Exclusion Criteria:

* co-infection with HIV or HBV
* previous treatment with peginterferon and/or ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving peginterferon alfa treatment at a medical centre
Sampling Method: Probability Sample
Enrollment: 2343 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (75):
- Belgium (21):
  - Aalst
  - Antwerp
  - Bruges
  - Brussels
  - Charleroi
  - Edegem
  - Genk
  - Ghent
  - Gilly (Charleroi)
  - Godinne
  - Haine-Saint-Paul
  - Kortrijk
  - Leuven
  - Liège
  - Namur
  - Ostend
  - Roeselare
  - Seraing
  - Sijsele
  - Tielt
  - Verviers
- Dublin, Ireland
- Italy (52):
  - Pescara, Abruzzo
  - Bisceglie, Apulia
  - Brindisi, Apulia
  - Casarano, Apulia
  - Castellana Grotte, Apulia
  - Foggia, Apulia
  - Galatina, Apulia
  - Taranto, Apulia
  - Catanzaro, Calabria
  - Vibo Valentia, Calabria
  - Barra, Campania
  - Benevento, Campania
  - Gragnano, Campania
  - Napoli, Campania
  - Nola, Campania
  - Bologna, Emilia-Romagna
  - Ferrara, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Basovizza (TS), Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Savona, Liguria
  - Brescia, Lombardy
  - Busto Arsizio, Lombardy
  - Cremona, Lombardy
  - Lecco, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Saronno, Lombardy
  - Treviglio, Lombardy
  - Isernia, Molise
  - Alessandria, Piedmont
  - Asti, Piedmont
  - Biella, Piedmont
  - Novara, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Catania, Sicily
  - Comiso, Sicily
  - Palermo, Sicily
  - Fermo, The Marches
  - Bolzano, Trentino-Alto Adige
  - Trento, Trentino-Alto Adige
  - Arezzo, Tuscany
  - Florence, Tuscany
  - Grosseto, Tuscany
  - Perugia, Umbria
  - Mestre (VE), Veneto
  - Padua, Veneto
  - Treviso, Veneto
  - Venezia, Veneto
  - Verona, Veneto
- London, United Kingdom

REFERENCES:
- [Derived] Ascione A, Bruno S, Coppola C, Mangia A, Orlandini A, Schmitz M, Deodato B, Puoti M. Treatment Outcomes and Predictors of Response in Treatment-Naive HCV Patients Treated with Peginterferon Alfa/Ribavirin in Real-World Italian Clinics: Sub-Analysis from the PROPHESYS Cohort. Hepatogastroenterology. 2014 Jun;61(132):1094-106. PMID 26158171
- [Derived] Ferenci P, Aires R, Ancuta I, Arohnson A, Cheinquer H, Delic D, Gschwantler M, Larrey D, Tallarico L, Schmitz M, Tatsch F, Ouzan D. A tool for selecting patients with a high probability of sustained virological response to peginterferon alfa-2a (40kD)/ribavirin. Liver Int. 2014 Nov;34(10):1550-9. doi: 10.1111/liv.12439. Epub 2014 Jan 9. PMID 24329937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2343 participants were enrolled in this study conducted from October 2007 to May 2011 at 125 centers in Belgium, Italy, United Kingdom, and Ireland.
Groups:
- Genotype 1 (G1): Eligible participants infected with hepatitis C virus (HCV) of Genotype 1 who received Pegasys® (Pegylated Interferon [PEG-IFN] alfa-2a) or PegIntron® (PEG-IFN alfa-2b) plus ribavirin dose according to the standard of care and in line with summary of product characteristics (SPCs)/local labeling for up to 72 weeks were observed.
- Genotype 2 (G2): Eligible participants infected with HCV of Genotype 2 who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 3 (G3): Eligible participants infected with HCV of Genotype 3 who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 4 (G4): Eligible participants infected with HCV of Genotype 4 who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 5/6 (G5/6): Eligible participants infected with HCV of Genotype 5/6 who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Unknown Genotype (UNK): Eligible participants infected with HCV of Genotype unknown who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
Period: Overall Study
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Started | 1128 | 572 | 484 | 143 | 11 | 5
Completed | 754 | 495 | 369 | 94 | 11 | 4
Not Completed | 374 | 77 | 115 | 49 | 0 | 1
Not completed — Death | 4 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 180 | 39 | 82 | 16 | 0 | 1
Not completed — Physician Decision | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 1 | 0 | 0 | 0
Not completed — Early Termination | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lab test not done | 7 | 0 | 0 | 1 | 0 | 0
Not completed — Miscellaneous | 4 | 5 | 6 | 0 | 0 | 0
Not completed — Non-responders | 104 | 5 | 11 | 25 | 0 | 0
Not completed — Other | 15 | 5 | 6 | 2 | 0 | 0
Not completed — Relapse | 20 | 8 | 2 | 3 | 0 | 0
Not completed — Result Not Available | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment Interrupted | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Treatment Never Started | 18 | 5 | 4 | 1 | 0 | 0
Not completed — Treatment Stopped | 2 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The all patient enrolled population included every participant for whom there was any data available in the PROPHESYS database.
Groups:
- Genotype 1 (G1): Eligible participants infected with HCV of Genotype 1 who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Total: Total of all reporting groups
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK) | Total
Number analyzed (Participants) | 1128 | 572 | 484 | 143 | 11 | 5 | 2343
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.52) | 54.2 (12.52) | 40.6 (9.20) | 46.6 (11.56) | 52.7 (12.82) | 51.4 (13.24) | 48.5 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532 | 291 | 134 | 53 | 4 | 3 | 1017
  Male | 596 | 281 | 350 | 90 | 7 | 2 | 1326

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population
Description: Sustained virological response (SVR) was defined as virological response (VR) at 24 weeks after end of treatment (EOT). Virological response was defined as hepatitis C virus ribonucleic acid (HCV RNA) of <15 international units per milliliter (IU/mL) as assessed by COBAS AmpliPrep/COBAS TaqMan (CAP/CTM) or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (lower limit of detection [LLOD] 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The SVR is reported in treatment naive HCV mono-infected modified all-treated (mTRT) population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN and ribavirin, and had at least one post-baseline HCV RNA result. Participants with a baseline (BL) result <50 IU/mL were excluded. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  PEG-IFN alfa-2a (n=778, 414, 353,114, 9, 2) | 46.1 [42.6 to 49.7] | 78.0 [73.7 to 81.9] | 68.3 [63.1 to 73.1] | 43.0 [33.7 to 52.6] | 55.6 [21.2 to 86.3] | 100.0 [15.8 to 100.0]
  PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 39.6 [32.4 to 47.1] | 81.7 [72.9 to 88.6] | 68.9 [57.1 to 79.2] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

2. Primary Outcome: Percentage of Participants With Sustained Virological Response by Type of Peginterferon and Genotype in Per Protocol Population
Description: Sustained virological response was defined as VR at 24 weeks after EOT. Virological response was defined as HCV RNA of <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The SVR is reported in treatment naive HCV mono-infected per protocol (PP) population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion and exclusion criteria of the study. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  PEG-IFN alfa-2a (n=704, 361, 299, 102, 7, 2) | 47.2 [43.4 to 50.9] | 79.5 [75.0 to 83.5] | 68.9 [63.3 to 74.1] | 40.2 [30.6 to 50.4] | 57.1 [18.4 to 90.1] | 100.0 [15.8 to 100.0]
  PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 39.2 [31.6 to 47.3] | 80.5 [70.6 to 88.2] | 69.1 [56.7 to 79.8] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

3. Secondary Outcome: Percentage of Participants With Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population Over Time
Description: Virological response (VR) was defined as HCV RNA <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The VR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN and ribavirin, and had at least one post-baseline HCV RNA result. Participants with a BL result <50 IU/mL were excluded. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 4.1 [2.8 to 5.8] | 21.7 [17.9 to 26.0] | 9.9 [7.0 to 13.5] | 2.6 [0.5 to 7.5] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 84.2]
  Wk2, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 3.8 [1.6 to 7.8] | 6.7 [2.7 to 13.4] | 6.8 [2.2 to 15.1] | 7.1 [0.2 to 33.9] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 25.6 [22.5 to 28.8] | 80.4 [76.3 to 84.1] | 70.8 [65.8 to 75.5] | 36.8 [28.0 to 46.4] | 44.4 [13.7 to 78.8] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 15.9 [10.9 to 22.1] | 75.0 [65.6 to 83.0] | 67.6 [55.7 to 78.0] | 42.9 [17.7 to 71.1] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 58.7 [55.2 to 62.2] | 91.8 [88.7 to 94.2] | 91.5 [88.1 to 94.2] | 66.7 [57.2 to 75.2] | 88.9 [51.8 to 99.7] | 50.0 [1.3 to 98.7]
  Wk12,PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 42.3 [35.0 to 49.8] | 91.3 [84.2 to 96.0] | 87.8 [78.2 to 94.3] | 50.0 [23.0 to 77.0] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  EOT, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 71.5 [68.2 to 74.6] | 91.3 [88.2 to 93.8] | 91.8 [88.4 to 94.4] | 66.7 [57.2 to 75.2] | 88.9 [51.8 to 99.7] | 100.0 [15.8 to 100.0]
  EOT, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 53.8 [46.3 to 61.2] | 90.4 [83.0 to 95.3] | 89.2 [79.8 to 95.2] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 84.2]
  12wk PEOT,PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 49.2 [45.7 to 52.8] | 80.0 [75.8 to 83.7] | 70.8 [65.8 to 75.5] | 46.5 [37.1 to 56.1] | 55.6 [21.2 to 86.3] | 100.0 [15.8 to 100.0]
  12wk PEOT, PEG-IFN alfa-2b (n=182,104, 4,14,2,2) | 40.7 [33.5 to 48.2] | 81.7 [72.9 to 88.6] | 70.3 [58.5 to 80.3] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

4. Secondary Outcome: Percentage of Participants With Virological Response by Type of Peginterferon and Genotype in Per Protocol Population Over Time
Description: Virological response (VR) was defined as HCV RNA <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The VR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 Weeks after EOT
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 4.0 [2.7 to 5.7] | 23.3 [19.0 to 28.0] | 10.4 [7.2 to 14.4] | 2.0 [0.2 to 6.9] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 84.2]
  Wk2, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 3.2 [1.0 to 7.2] | 8.0 [3.3 to 15.9] | 7.4 [2.4 to 16.3] | 7.1 [0.2 to 33.9] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=704,361,299,102,7, 2) | 26.4 [23.2 to 29.8] | 82.5 [78.2 to 86.3] | 71.2 [65.7 to 76.3] | 38.2 [28.8 to 48.4] | 28.6 [3.7 to 71.0] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 15.2 [10.0 to 21.8] | 75.9 [65.5 to 84.4] | 64.7 [52.2 to 75.9] | 42.9 [17.7 to 71.1] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=704,361,299,102,7, 2) | 59.9 [56.2 to 63.6] | 93.1 [89.9 to 95.5] | 92.3 [88.7 to 95.1] | 68.6 [58.7 to 77.5] | 85.7 [42.1 to 99.6] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 42.4 [34.6 to 50.5] | 92.0 [84.1 to 96.7] | 86.8 [76.4 to 93.8] | 50.0 [23.0 to 77.0] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  EOT, PEG-IFN alfa-2a (n=704,361,299,102, 7, 2) | 72.9 [69.4 to 76.1] | 92.2 [89.0 to 94.8] | 92.3 [88.7 to 95.1] | 65.7 [55.6 to 74.8] | 85.7 [42.1 to 99.6] | 100.0 [15.8 to 100.0]
  EOT, PEG-IFN alfa-2b (n=158, 87, 68,14, 2, 2) | 52.5 [44.4 to 60.5] | 89.7 [81.3 to 95.2] | 89.7 [79.9 to 95.8] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 84.2]
  12wk PEOT,PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 50.3 [46.5 to 54.0] | 81.4 [77.0 to 85.3] | 71.2 [65.7 to 76.3] | 44.1 [34.3 to 54.3] | 57.1 [18.4 to 90.1] | 100.0 [15.8 to 100.0]
  12wk PEOT, PEG-IFN alfa-2b (n=158, 87, 68,14,2,2) | 39.9 [32.2 to 48.0] | 80.5 [70.6 to 88.2] | 70.6 [58.3 to 81.0] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

5. Secondary Outcome: Percentage of Participants With Modified Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population Over Time
Description: Modified virological response (mVR) was defined as HCV RNA <50 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The mVR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 Weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 4.8 [3.4 to 6.5] | 24.9 [20.8 to 29.3] | 12.7 [9.5 to 16.7] | 3.5 [1.0 to 8.7] | 0.0 [0.0 to 33.6] | 50.0 [1.3 to 98.7]
  Wk2, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 3.8 [1.6 to 7.8] | 10.6 [5.4 to 18.1] | 12.2 [5.7 to 21.8] | 7.1 [0.2 to 33.9] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 30.5 [27.2 to 33.8] | 85.5 [81.7 to 88.8] | 75.1 [70.2 to 79.5] | 41.2 [32.1 to 50.8] | 44.4 [13.7 to 78.8] | 100.0 [15.8 to 100.0]
  Wk4, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 20.9 [15.2 to 27.5] | 86.5 [78.4 to 92.4] | 74.3 [62.8 to 83.8] | 42.9 [17.7 to 71.1] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 63.6 [60.1 to 67.0] | 94.0 [91.2 to 96.1] | 93.2 [90.1 to 95.6] | 70.2 [60.9 to 78.4] | 100.0 [66.4 to 100.0] | 100.0 [15.8 to 100.0]
  Wk12, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 47.8 [40.4 to 55.3] | 94.2 [87.9 to 97.9] | 93.2 [84.9 to 97.8] | 50.0 [23.0 to 77.0] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  EOT, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 73.8 [70.5 to 76.8] | 92.8 [89.8 to 95.1] | 92.4 [89.1 to 94.9] | 67.5 [58.1 to 76.0] | 88.9 [51.8 to 99.7] | 100.0 [15.8 to 100.0]
  EOT, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 57.1 [49.6 to 64.4] | 92.3 [85.4 to 96.6] | 89.2 [79.8 to 95.2] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 84.2]
  12wk PEOT, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 50.0 [46.4 to 53.6] | 80.2 [76.0 to 83.9] | 71.4 [66.4 to 76.0] | 46.5 [37.1 to 56.1] | 66.7 [29.9 to 92.5] | 100.0 [15.8 to 100.0]
  12wk PEOT, PEG-IFN alfa-2b (n=182,104, 4,14,2,2) | 40.7 [33.5 to 48.2] | 83.7 [75.1 to 90.2] | 70.3 [58.5 to 80.3] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

6. Secondary Outcome: Percentage of Participants With Modified Virological Response Over Time by Type of Peginterferon and Genotype in Per Protocol Population Over Time
Description: Modified virological response (mVR) is defined as HCV RNA <50 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The mVR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 Weeks after EOT
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=704,361,299,102,7, 2) | 4.7 [3.2 to 6.5] | 26.0 [21.6 to 30.9] | 12.7 [9.2 to 17.0] | 2.9 [0.6 to 8.4] | 0.0 [0.0 to 41.0] | 50.0 [1.3 to 98.7]
  Wk2, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 3.2 [1.0 to 7.2] | 12.6 [6.5 to 21.5] | 13.2 [6.2 to 23.6] | 7.1 [0.2 to 33.9] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=704, 361,299,102,7,2) | 31.7 [28.3 to 35.3] | 87.3 [83.4 to 90.5] | 74.9 [69.6 to 79.7] | 43.1 [33.4 to 53.3] | 28.6 [3.7 to 71.0] | 100.0 [15.8 to 100.0]
  Wk4, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 20.9 [14.8 to 28.1] | 88.5 [79.9 to 94.3] | 72.1 [59.9 to 82.3] | 42.9 [17.7 to 71.1] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 65.1 [61.4 to 68.6] | 95.0 [92.2 to 97.0] | 94.0 [90.7 to 96.4] | 71.6 [61.8 to 80.1] | 100.0 [59.0 to 100.0] | 100.0 [15.8 to 100.0]
  Wk12,PEG-IFN alfa-2b (n=158, 87, 68,14, 2, 2) | 48.1 [40.1 to 56.2] | 94.3 [87.1 to 98.1] | 92.6 [83.7 to 97.6] | 50.0 [23.0 to 77.0] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  EOT, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 74.9 [71.5 to 78.0] | 93.6 [90.6 to 95.9] | 92.6 [89.1 to 95.3] | 66.7 [56.6 to 75.7] | 85.7 [42.1 to 99.6] | 100.0 [15.8 to 100.0]
  EOT, PEG-IFN alfa-2b (n=158, 87, 68,14, 2, 2) | 56.3 [48.2 to 64.2] | 92.0 [84.1 to 96.7] | 89.7 [79.9 to 95.8] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 84.2]
  12wk PEOT, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 51.1 [47.4 to 54.9] | 81.4 [77.0 to 85.3] | 71.9 [66.4 to 76.9] | 44.1 [34.3 to 54.3] | 57.1 [18.4 to 90.1] | 100.0 [15.8 to 100.0]
  12wk PEOT, PEG-IFN alfa-2b (n=158,87,68,14,2,2) | 39.9 [32.2 to 48.0] | 82.8 [73.2 to 90.0] | 70.6 [58.3 to 81.0] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

7. Primary Outcome: Percentage of Participants With Modified Sustained Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population
Description: Modified sustained virological response (mSVR) was defined as modified virological response (mVR) of HCV RNA <50 IU/mL at 24 weeks after EOT. The mSVR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  PEG-IFN alfa-2a (n=778, 414, 353,114, 9, 2) | 46.5 [43.0 to 50.1] | 78.3 [74.0 to 82.1] | 68.6 [63.4 to 73.4] | 43.0 [33.7 to 52.6] | 66.7 [29.9 to 92.5] | 100.0 [15.8 to 100.0]
  PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 39.6 [32.4 to 47.1] | 82.7 [74.0 to 89.4] | 68.9 [57.1 to 79.2] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]
Statistical Analysis 1: Comparison: Genotype 1 (G1); The statistical analysis is presented for Gamma-Glutamyl Transferase (Gamma-GT) in log10 international units per liter (IU/L) at BL. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week [Wk]12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0211, Regression, Logistic; Odds Ratio (OR) = 0.527, 95% CI 2-sided [0.306 to 0.908]
Statistical Analysis 2: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.078, 95% CI 2-sided [1.065 to 1.092]
Statistical Analysis 3: Comparison: Genotype 1 (G1); The statistical analysis is presented for cumulative ribavirin dose per 10000 mg, during the first 12 weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0053, Regression, Logistic; Odds Ratio (OR) = 1.220, 95% CI 2-sided [1.061 to 1.403]
Statistical Analysis 4: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (< 140 vs >=180). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0079, Regression, Logistic; Odds Ratio (OR) = 0.464, 95% CI 2-sided [0.264 to 0.818]
Statistical Analysis 5: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (>=140 - < 180 vs >=180). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.1808, Regression, Logistic; Odds Ratio (OR) = 0.737, 95% CI 2-sided [0.471 to 1.153]
Statistical Analysis 6: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.082, 95% CI 2-sided [1.069 to 1.095]
Statistical Analysis 7: Comparison: Genotype 2 (G2); The statistical analysis is presented for Weight per 10 kilogram (kg). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 0.676, 95% CI 2-sided [0.542 to 0.844]
Statistical Analysis 8: Comparison: Genotype 2 (G2); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0041, Regression, Logistic; Odds Ratio (OR) = 0.573, 95% CI 2-sided [0.392 to 0.838]
Statistical Analysis 9: Comparison: Genotype 2 (G2); [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.094, 95% CI 2-sided [1.048 to 1.142]
Statistical Analysis 10: Comparison: Genotype 2 (G2); The statistical analysis is presented for cumulative PEG-IFN alfa-2a dose per 1000 ug, first 12 weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0031, Regression, Logistic; Odds Ratio (OR) = 7.945, 95% CI 2-sided [2.013 to 31.359]
Statistical Analysis 11: Comparison: Genotype 2 (G2); The statistical analysis is presented for body mass index (BMI) in kilogram per square meter (kg/m^2). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 0.900, 95% CI 2-sided [0.844 to 0.959]
Statistical Analysis 12: Comparison: Genotype 2 (G2); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0085, Regression, Logistic; Odds Ratio (OR) = 0.619, 95% CI 2-sided [0.433 to 0.885]
Statistical Analysis 13: Comparison: Genotype 2 (G2); [analysis description as in outcome 7, analysis 6]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.130, 95% CI 2-sided [1.087 to 1.174]
Statistical Analysis 14: Comparison: Genotype 3 (G3); The statistical analysis is presented for Weight per 10 kg. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0341, Regression, Logistic; Odds Ratio (OR) = 0.784, 95% CI 2-sided [0.626 to 0.982]
Statistical Analysis 15: Comparison: Genotype 3 (G3); The statistical analysis is presented for aspartate aminotransferase (AST) ratio at BL (> 1.5 vs <=1.5). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0443, Regression, Logistic; Odds Ratio (OR) = 0.575, 95% CI 2-sided [0.335 to 0.986]
Statistical Analysis 16: Comparison: Genotype 3 (G3); [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.100, 95% CI 2-sided [1.057 to 1.144]
Statistical Analysis 17: Comparison: Genotype 3 (G3); The statistical analysis is presented for cumulative PEG-IFN alfa-2a dose per 1000 ug, during the first 12 weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0039, Regression, Logistic; Odds Ratio (OR) = 22.867, 95% CI 2-sided [2.730 to 191.56]
Statistical Analysis 18: Comparison: Genotype 3 (G3); The statistical analysis is presented for Weight per 10 kg. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0244, Regression, Logistic; Odds Ratio (OR) = 0.780, 95% CI 2-sided [0.628 to 0.968]
Statistical Analysis 19: Comparison: Genotype 3 (G3); [analysis description as in outcome 7, analysis 6]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.128, 95% CI 2-sided [1.086 to 1.172]
Statistical Analysis 20: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0453, Regression, Logistic; Odds Ratio (OR) = 0.547, 95% CI 2-sided [0.303 to 0.987]
Statistical Analysis 21: Comparison: Genotype 1 (G1); The statistical analysis is presented for Gamma-GT in log10 (IU/L) at BL. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0184, Regression, Logistic; Odds Ratio (OR) = 0.133, 95% CI 2-sided [0.025 to 0.712]
Statistical Analysis 22: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in Weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.103, 95% CI 2-sided [1.072 to 1.134]
Statistical Analysis 23: Comparison: Genotype 1 (G1); The statistical analysis is presented for weight per 10 kg. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 0.543, 95% CI 2-sided [0.370 to 0.798]
Statistical Analysis 24: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0017, Regression, Logistic; Odds Ratio (OR) = 0.359, 95% CI 2-sided [0.189 to 0.679]
Statistical Analysis 25: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.080, 95% CI 2-sided [1.047 to 1.114]
Statistical Analysis 26: Comparison: Genotype 1 (G1); The statistical analysis is presented for cumulative ribavirin dose per 10000 mg. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0042, Regression, Logistic; Odds Ratio (OR) = 1.093, 95% CI 2-sided [1.029 to 1.162]
Statistical Analysis 27: Comparison: Genotype 1 (G1); The statistical analysis is presented for Gamma-GT in log10 (IU/L) at BL. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0168, Regression, Logistic; Odds Ratio (OR) = 0.535, 95% CI 2-sided [0.320 to 0.893]
Statistical Analysis 28: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (< 140 vs >=180). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0128, Regression, Logistic; Odds Ratio (OR) = 0.501, 95% CI 2-sided [0.291 to 0.864]
Statistical Analysis 29: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (>=140 - < 180 vs >=180). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.4634, Regression, Logistic; Odds Ratio (OR) = 0.853, 95% CI 2-sided [0.558 to 1.305]
Statistical Analysis 30: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (Rapid Virological Response [RVR] vs No RVR/EVR [Early Virological Response]). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 19.655, 95% CI 2-sided [9.725 to 39.722]
Statistical Analysis 31: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (cEVR [Complete Early Virological Response] vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 8.569, 95% CI 2-sided [4.408 to 16.658]
Statistical Analysis 32: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (pEVR [Partial Early Virological Response] vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0089, Regression, Logistic; Odds Ratio (OR) = 2.519, 95% CI 2-sided [1.260 to 5.034]
Statistical Analysis 33: Comparison: Genotype 2 (G2); The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0037, Regression, Logistic; Odds Ratio (OR) = 0.908, 95% CI 2-sided [0.851 to 0.969]
Statistical Analysis 34: Comparison: Genotype 2 (G2); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 0.553, 95% CI 2-sided [0.379 to 0.805]
Statistical Analysis 35: Comparison: Genotype 2 (G2); The statistical analysis is presented for On-treatment response (RVR vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 16.537, 95% CI 2-sided [3.654 to 74.849]
Statistical Analysis 36: Comparison: Genotype 2 (G2); The statistical analysis is presented for on-treatment response (cEVR vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0733, Regression, Logistic; Odds Ratio (OR) = 4.386, 95% CI 2-sided [0.870 to 22.114]
Statistical Analysis 37: Comparison: Genotype 2 (G2); The statistical analysis is presented for on-treatment response (pEVR vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.3478, Regression, Logistic; Odds Ratio (OR) = 2.352, 95% CI 2-sided [0.394 to 14.031]
Statistical Analysis 38: Comparison: Genotype 3 (G3); The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0264, Regression, Logistic; Odds Ratio (OR) = 0.729, 95% CI 2-sided [0.552 to 0.964]
Statistical Analysis 39: Comparison: Genotype 3 (G3); [analysis description as in outcome 7, analysis 35]; Test type: Superiority or Other; p = 0.0096, Regression, Logistic; Odds Ratio (OR) = 6.658, 95% CI 2-sided [1.586 to 27.946]
Statistical Analysis 40: Comparison: Genotype 3 (G3); [analysis description as in outcome 7, analysis 36]; Test type: Superiority or Other; p = 0.0421, Regression, Logistic; Odds Ratio (OR) = 4.734, 95% CI 2-sided [1.057 to 21.203]
Statistical Analysis 41: Comparison: Genotype 3 (G3); [analysis description as in outcome 7, analysis 37]; Test type: Superiority or Other; p = 0.6004, Regression, Logistic; Odds Ratio (OR) = 0.602, 95% CI 2-sided [0.090 to 4.014]
Statistical Analysis 42: Comparison: Genotype 1 (G1); The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0418, Regression, Logistic; Odds Ratio (OR) = 0.715, 95% CI 2-sided [0.517 to 0.988]
Statistical Analysis 43: Comparison: Genotype 1 (G1); The statistical analysis is presented for Gamma-GT in log10 (IU/L) at BL. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0279, Regression, Logistic; Odds Ratio (OR) = 0.198, 95% CI 2-sided [0.047 to 0.839]
Statistical Analysis 44: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (RVR vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 40.880, 95% CI 2-sided [7.474 to 223.61]
Statistical Analysis 45: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (cEVR vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 42.395, 95% CI 2-sided [8.724 to 206.02]
Statistical Analysis 46: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (pEVR vs No RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0087, Regression, Logistic; Odds Ratio (OR) = 8.247, 95% CI 2-sided [1.704 to 39.908]

8. Primary Outcome: Percentage of Participants With Modified Sustained Virological Response by Type of Peginterferon and Genotype in Per Protocol Population
Description: Modified sustained virological response is defined as mVR of HCV RNA <50 IU/mL at 24 weeks after EOT. The mSVR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  PEG-IFN alfa-2a (n=704, 361, 299, 102, 7, 2) | 47.6 [43.8 to 51.3] | 79.5 [75.0 to 83.5] | 69.2 [63.7 to 74.4] | 40.2 [30.6 to 50.4] | 57.1 [18.4 to 90.1] | 100.0 [15.8 to 100.0]
  PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 39.2 [31.6 to 47.3] | 81.6 [71.9 to 89.1] | 69.1 [56.7 to 79.8] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 84.2]

9. Secondary Outcome: Percentage of Participants With at Least a 2-logarithm10 Drop in Hepatitis C Virus Ribonucleic Acid in Modified All Treated Population at Week 2, Week 4 and Week 12
Description: Participants with 2-logarithm (log) drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 2 log drop in HCV RNA was defined as drop of HCV viral load by 99%. The 2 log drop in HCV RNA is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 14.4 [12.0 to 17.1] | 33.8 [29.3 to 38.6] | 20.1 [16.1 to 24.7] | 5.3 [2.0 to 11.1] | 0.0 [0.0 to 33.6] | 50.0 [1.3 to 98.7]
  Wk2, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 10.4 [6.4 to 15.8] | 24.0 [16.2 to 33.4] | 20.3 [11.8 to 31.2] | 14.3 [1.8 to 42.8] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 59.0 [55.4 to 62.5] | 90.8 [87.6 to 93.4] | 85.0 [80.8 to 88.5] | 64.0 [54.5 to 72.8] | 66.7 [29.9 to 92.5] | 100.0 [15.8 to 100.0]
  Wk4, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 46.2 [38.8 to 53.7] | 94.2 [87.9 to 97.9] | 85.1 [75.0 to 92.3] | 42.9 [17.7 to 71.1] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 83.4 [80.6 to 86.0] | 96.1 [93.8 to 97.8] | 96.0 [93.4 to 97.8] | 77.2 [68.4 to 84.5] | 100.0 [66.4 to 100.0] | 100.0 [15.8 to 100.0]
  Wk12, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 73.1 [66.0 to 79.4] | 99.0 [94.8 to 100.0] | 97.3 [90.6 to 99.7] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]

10. Secondary Outcome: Percentage of Participants With at Least a 2-logarithm10 Drop in Hepatitis C Virus Ribonucleic Acid in Per Protocol Population at Week 2, Week 4 and Week 12
Description: Participants with 2-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 2 log drop in HCV RNA was defined as drop of HCV viral load by 99%. The 2 log drop in HCV RNA is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 14.5 [12.0 to 17.3] | 36.0 [31.1 to 41.2] | 20.4 [16.0 to 25.4] | 4.9 [1.6 to 11.1] | 0.0 [0.0 to 41.0] | 50.0 [1.3 to 98.7]
  Wk2, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 10.1 [5.9 to 15.9] | 26.4 [17.6 to 37.0] | 22.1 [12.9 to 33.8] | 14.3 [1.8 to 42.8] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 59.9 [56.2 to 63.6] | 92.5 [89.3 to 95.0] | 84.9 [80.4 to 88.8] | 65.7 [55.6 to 74.8] | 57.1 [18.4 to 90.1] | 100.0 [15.8 to 100.0]
  Wk4, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 45.6 [37.6 to 53.7] | 95.4 [88.6 to 98.7] | 83.8 [72.9 to 91.6] | 42.9 [17.7 to 71.1] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 84.8 [81.9 to 87.4] | 96.7 [94.3 to 98.3] | 96.7 [93.9 to 98.4] | 78.4 [69.2 to 86.0] | 100.0 [59.0 to 100.0] | 100.0 [15.8 to 100.0]
  Wk12,PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 73.4 [65.8 to 80.1] | 98.9 [93.8 to 100.0] | 97.1 [89.8 to 99.6] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]

11. Secondary Outcome: Percentage of Participants With at Least a 1-logarithm10 Drop in Hepatitis C Virus Ribonucleic Acid in Modified All Treated Population at Week 2, Week 4 and Week 12
Description: Participants with 1-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 1- log drop in HCV RNA was defined as drop of HCV viral load by 90%. The 1- log drop in HCV RNA was reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 23.7 [20.7 to 26.8] | 37.2 [32.5 to 42.1] | 21.8 [17.6 to 26.5] | 8.8 [4.3 to 15.5] | 0.0 [0.0 to 33.6] | 50.0 [1.3 to 98.7]
  Wk2, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 18.7 [13.3 to 25.1] | 26.9 [18.7 to 36.5] | 24.3 [15.1 to 35.7] | 21.4 [4.7 to 50.8] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 79.6 [76.6 to 82.3] | 93.0 [90.1 to 95.3] | 87.8 [83.9 to 91.0] | 78.1 [69.4 to 85.3] | 88.9 [51.8 to 99.7] | 100.0 [15.8 to 100.0]
  Wk4, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 75.8 [68.9 to 81.9] | 96.2 [90.4 to 98.9] | 89.2 [79.8 to 95.2] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 93.6 [91.6 to 95.2] | 98.1 [96.2 to 99.2] | 97.2 [94.9 to 98.6] | 86.0 [78.2 to 91.8] | 100.0 [66.4 to 100.0] | 100.0 [15.8 to 100.0]
  Wk12, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 89.0 [83.5 to 93.2] | 99.0 [94.8 to 100.0] | 98.6 [92.7 to 100.0] | 78.6 [49.2 to 95.3] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]

12. Primary Outcome: Percentage of Participants With Predictive Values of Virological Response on Modified Sustained Virological Response After Treatment Initiation in Modified All Treated Population
Description: The probability that a participant who developed VR by Week 4 and 12 and also achieved mSVR at 24 weeks after EOT was called the positive predictive value (PPV) of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the negative predictive value (NPV) of the VR by Wk 4 and 12 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected mTRT participants who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  Wk4,PEG-IFN alfa-2a, PPV (n=733,397,325,104,8,2) | 74.9 [68.3 to 80.7] | 84.7 [80.4 to 88.4] | 74.8 [68.9 to 80.1] | 64.3 [48.0 to 78.4] | 100.0 [39.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, PEG-IFN alfa-2a, NPV (n=733,397,325,104,8,2) | 64.0 [59.8 to 68.1] | 51.6 [38.7 to 64.2] | 52.0 [40.2 to 63.7] | 71.0 [58.1 to 81.8] | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5]
  Wk4, PEG-IFN alfa-2b, PPV (n=177,101,71,14,2,2) | 72.4 [52.8 to 87.3] | 91.0 [82.4 to 96.3] | 80.0 [66.3 to 90.0] | 66.7 [22.3 to 95.7] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, PEG-IFN alfa-2b, NPV (n=177,101,71,14,2,2) | 67.6 [59.4 to 75.0] | 47.8 [26.8 to 69.4] | 61.9 [38.4 to 81.9] | 87.5 [47.3 to 99.7] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,PEG-IFN alfa-2a,PPV (n=768,412,350,109,9,2) | 64.6 [60.0 to 68.9] | 81.8 [77.6 to 85.6] | 72.4 [67.2 to 77.2] | 59.2 [47.3 to 70.4] | 75.0 [34.9 to 96.8] | 100.0 [2.5 to 100.0]
  Wk12,PEG-IFN alfa-2a, NPV(n=768,412,350,109,9,2) | 80.1 [75.2 to 84.4] | 59.4 [40.6 to 76.3] | 74.1 [53.7 to 88.9] | 93.9 [79.8 to 99.3] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12,PEG-IFN alfa-2b, PPV (n=181, 104,74,14,2,2) | 68.8 [57.3 to 78.9] | 86.3 [77.7 to 92.5] | 73.8 [61.5 to 84.0] | 71.4 [29.0 to 96.3] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, PEG-IFN alfa-2b, NPV (n=181, 104,74,14,2,2) | 81.7 [72.9 to 88.6] | 55.6 [21.2 to 86.3] | 66.7 [29.9 to 92.5] | 100.0 [59.0 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0]

13. Primary Outcome: Percentage of Participants With Predictive Values of Virological Response on Modified Sustained Virological Response After Treatment Initiation in Per Protocol Population
Description: The probability that a participant who developed VR by Week 4 and 12 and also achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 4 and 12 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  Wk4,PEG-IFN alfa-2a, PPV (n=668,351,275,93,6,2) | 75.8 [69.0 to 81.8] | 85.6 [81.1 to 89.4] | 73.7 [67.3 to 79.5] | 61.5 [44.6 to 76.6] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4,PEG-IFN alfa-2a, NPV (n=668,351,275,93,6,2) | 63.5 [59.0 to 67.8] | 49.1 [35.1 to 63.2] | 45.2 [32.5 to 58.3] | 74.1 [60.3 to 85.0] | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5]
  Wk4, PEG-IFN alfa-2b, PPV (n=155,85,65,14,2,2) | 75.0 [53.3 to 90.2] | 90.9 [81.3 to 96.6] | 81.8 [67.3 to 91.8] | 66.7 [22.3 to 95.7] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, PEG-IFN alfa-2b, NPV (n=155,85,65,14,2,2) | 68.7 [60.0 to 76.5] | 52.6 [28.9 to 75.6] | 61.9 [38.4 to 81.9] | 87.5 [47.3 to 99.7] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,PEG-IFN alfa-2a, PPV(n=697,359,296,98,7,2) | 65.2 [60.4 to 69.7] | 82.4 [77.9 to 86.4] | 72.5 [66.8 to 77.6] | 55.7 [43.3 to 67.6] | 66.7 [22.3 to 95.7] | 100.0 [2.5 to 100.0]
  Wk12,PEG-IFN alfa-2a, NPV (n=697,359,296,98,7,2) | 79.6 [74.4 to 84.2] | 56.5 [34.5 to 76.8] | 70.0 [45.7 to 88.1] | 96.4 [81.7 to 99.9] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, PEG-IFN alfa-2b, PPV (n=158, 87,68,14,2,2) | 68.7 [56.2 to 79.4] | 85.0 [75.3 to 92.0] | 74.6 [61.6 to 85.0] | 71.4 [29.0 to 96.3] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, PEG-IFN alfa-2b, NPV (n=158, 87,68,14,2,2) | 82.4 [73.0 to 89.6] | 57.1 [18.4 to 90.1] | 66.7 [29.9 to 92.5] | 100.0 [59.0 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0]

14. Secondary Outcome: Percentage of Participants With at Least a 1-logarithm 10 Drop in Hepatitis C Virus Ribonucleic Acid in Per Protocol Population at Week 2, Week 4 and Week 12
Description: Participants with 1-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 1- log drop in HCV RNA was defined as drop of HCV viral load by 90%. The 1- log drop in HCV RNA was reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 24.0 [20.9 to 27.3] | 39.9 [34.8 to 45.1] | 22.4 [17.8 to 27.6] | 7.8 [3.4 to 14.9] | 0.0 [0.0 to 41.0] | 50.0 [1.3 to 98.7]
  Wk2,PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 17.1 [11.6 to 23.9] | 28.7 [19.5 to 39.4] | 26.5 [16.5 to 38.6] | 21.4 [4.7 to 50.8] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
  Wk4, PEG-IFN alfa-2a (n=704,361,299,102,7, 2) | 81.3 [78.2 to 84.1] | 94.7 [91.9 to 96.8] | 88.3 [84.1 to 91.7] | 79.4 [70.3 to 86.8] | 85.7 [42.1 to 99.6] | 100.0 [15.8 to 100.0]
  Wk4, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 76.6 [69.2 to 82.9] | 96.6 [90.3 to 99.3] | 88.2 [78.1 to 94.8] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]
  Wk12, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 94.9 [93.0 to 96.4] | 98.3 [96.4 to 99.4] | 98.0 [95.7 to 99.3] | 87.3 [79.2 to 93.0] | 100.0 [59.0 to 100.0] | 100.0 [15.8 to 100.0]
  Wk12, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 90.5 [84.8 to 94.6] | 98.9 [93.8 to 100.0] | 98.5 [92.1 to 100.0] | 78.6 [49.2 to 95.3] | 100.0 [15.8 to 100.0] | 50.0 [1.3 to 98.7]

15. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response on Modified Sustained Virological Response After Treatment Initiation in Modified All Treated Population
Description: The probability that a participant who developed VR by Wk 2 achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 4 and 12 for mSVR. Predictive Values of VR was reported in treatment naive HCV mono-infected mTRT population participants who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: 24 weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a, PPV (n=267,174,98,16,0, 1) | 84.4 [67.2 to 94.7] | 92.2 [84.6 to 96.8] | 77.1 [59.9 to 89.6] | 33.3 [0.8 to 90.6] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk2, PEG-IFN alfa-2a,NPV (n=267, 174,98,16, 0, 1) | 51.9 [45.3 to 58.5] | 22.6 [14.2 to 33.0] | 28.6 [17.9 to 41.3] | 69.2 [38.6 to 90.9] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | 0.0 [0.0 to 97.5]
  Wk2, PEG-IFN alfa-2b, PPV (n=54, 29, 19,7,1,1) | 57.1 [18.4 to 90.1] | 71.4 [29.0 to 96.3] | 60.0 [14.7 to 94.7] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk2, PEG-IFN alfa-2b, NPV (n=54,29,19,7,1, 1) | 59.6 [44.3 to 73.6] | 13.6 [2.9 to 34.9] | 28.6 [8.4 to 58.1] | 50.0 [11.8 to 88.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.

16. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response on Modified Sustained Virological Response After Treatment Initiation in Per Protocol Population
Description: The probability that a participant who developed VR by Wk 2 and achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 2 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 2 for mSVR. Predictive values of VR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: 24 weeks after EOT
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  Wk2, PEG-IFN alfa-2a, PPV (n=246, 63,87,14,0,1) | 82.1 [63.1 to 93.9] | 92.9 [85.1 to 97.3] | 74.2 [55.4 to 88.1] | 0.0 [0.0 to 84.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk2, PEG-IFN alfa-2a, NPV (n=246, 163,87,14,0,1) | 51.8 [45.0 to 58.6] | 21.5 [13.1 to 32.2] | 28.6 [17.3 to 42.2] | 75.0 [42.8 to 94.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | 0.0 [0.0 to 97.5]
  Wk2, PEG-IFN alfa-2b, PPV (n=43, 26,19,7,1,1) | 60.0 [14.7 to 94.7] | 71.4 [29.0 to 96.3] | 60.0 [14.7 to 94.7] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk2, PEG-IFN alfa-2b, NPV (n=43, 26,19,7,1,1) | 55.3 [38.3 to 71.4] | 15.8 [3.4 to 39.6] | 28.6 [8.4 to 58.1] | 50.0 [11.8 to 88.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.

17. Secondary Outcome: Number of Participants With Response by Disjoint Categories in Modified All-Treated Population at Week 4 and Week 12
Description: Rapid virological response (RVR) was defined as VR by Wk 4, Modified rapid virological response (mRVR) was defined as mVR by Wk 4, complete early virological response (cEVR) was defined as VR by Wk 12, but no RVR, modified complete early virological response (mcEVR) was defined as mVR by Wk 12, but no mRVR, partial early virological response (pEVR) was defined as at least a 2-log10 drop in HCV RNA as compared to baseline (including HCV RNA values <50 IU/mL) by, Wk 12, but no RVR and no cEVR, modified partial early virological response (mpEVR) was defined as at least a 2-log10 drop in HCV RNA as compared to baseline by Wk 12, but no mRVR and no mcEVR. The data is reported in treatment naive HCV mono-infected mTRT participants who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: number of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
number of participants
  RVR, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 199 | 333 | 250 | 42 | 4 | 1
  RVR, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 29 | 78 | 50 | 6 | 1 | 1
  mRVR,PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 237 | 354 | 265 | 47 | 4 | 2
  mRVR, PEG-IFN alfa-2b (n=182, 104,74,14, 2, 2) | 38 | 90 | 55 | 6 | 1 | 1
  cEVR, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 258 | 47 | 73 | 34 | 4 | 0
  cEVR, PEG-IFN alfa-2b (n=182, 104, 74,14, 2, 2) | 48 | 17 | 15 | 1 | 0 | 0
  mcEVR, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 258 | 35 | 64 | 33 | 5 | 0
  mCEVR, PEG-IFN alfa-2b (n=182,104,74,14,2, 2) | 49 | 8 | 14 | 1 | 0 | 0
  pEVR, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 192 | 18 | 16 | 12 | 1 | 1
  pEVR, PEG-IFN alfa-2b (n=182, 104,74,14, 2, 2) | 56 | 8 | 7 | 1 | 1 | 0
  mpEVR, PEG-IFN alfa-2a (n=778,414,353,114,9,2) | 154 | 9 | 10 | 8 | 0 | 0
  mpEVR, PEG-IFN alfa-2b (n=182,104, 74,14,2, 2) | 46 | 5 | 3 | 1 | 1 | 0

18. Secondary Outcome: Number of Participants With Response by Disjoint Categories in Per-Protocol Population at Week 4 and Week 12
Description: RVR was defined as as VR by Wk 4, mRVR was defined as mVR by Wk 4, cEVR was defined as VR by Wk 12, but no RVR, mcEVR was defined as mVR by Wk 12, but no mRVR, pEVR was defined as at least a 2-log10 drop in HCV RNA as compared to baseline (including HCV RNA values <50 IU/mL) by Wk 12, but no RVR and no cEVR, mpEVR was defined as at least a 2-log10 drop in HCV RNA as compared to baseline by Wk 12, but no mRVR and no mcEVR. The data is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
number of participants
  RVR, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 186 | 298 | 213 | 39 | 2 | 1
  RVR, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 24 | 66 | 44 | 6 | 1 | 1
  mRVR, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 223 | 315 | 224 | 44 | 2 | 2
  mRVR, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 33 | 77 | 49 | 6 | 1 | 1
  cEVR, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 236 | 38 | 63 | 31 | 4 | 0
  cEVR, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 43 | 14 | 15 | 1 | 0 | 0
  mcEVR, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 235 | 28 | 57 | 29 | 5 | 0
  mCEVR, PEG-IFN alfa-2b (n=158, 87, 68,14, 2, 2) | 43 | 5 | 14 | 1 | 0 | 0
  pEVR, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 175 | 13 | 13 | 10 | 1 | 1
  pEVR, PEG-IFN alfa-2b (n=158, 87, 68, 14, 2, 2) | 49 | 6 | 7 | 1 | 1 | 0
  mpEVR, PEG-IFN alfa-2a (n=704,361,299,102,7,2) | 139 | 6 | 8 | 7 | 0 | 0
  mpEVR, PEG-IFN alfa-2b (n=158, 87, 68,14, 2, 2) | 40 | 4 | 3 | 1 | 1 | 0

19. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Modified All-Treated Population at 12 Weeks After End of Treatment
Description: Participants whose last test result in their respective follow-up time window showed mVR were considered to have maintained their modified end of treatment response (mEOT-R). Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The number of participants with relapse was reported in treatment naive mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 12 weeks after EOT
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  12wk PEOT, PEG-IFN alfa-2a (n=257,193,109,14,0,0) | 30.0 | 10.9 | 14.7 | 21.4 | 0 | 0
  12wk PEOT, PEG-IFN alfa-2b (n=36,50,27,3,0,0) | 22.2 | 4.0 | 7.4 | 33.3 | 0 | 0

20. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Per Protocol Population at 12 Weeks After End of Treatment
Description: Participants whose last test result in their respective follow-up time window showed mVR were considered to have maintained their mEOT-R. Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The number of participants with relapse was reported in treatment naive PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 12 weeks after EOT
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Genotype 1 (G1): Eligible participants infected with HCV inclusive of all Genotypes who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  12Wk PEOT, PEG-IFN alfa-2a (n=239,175,98,12,0,0) | 29.3 | 10.3 | 14.3 | 25.0 | 0 | 0
  12wk PEOT, PEG-IFN alfa-2b (n=28,43,25,3,0,0) | 25.0 | 4.7 | 8.0 | 33.3 | 0 | 0

21. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Modified All-Treated Population at 24 Weeks After End of Treatment
Description: Participants whose last test result in the follow-up time window showed mVR were considered to have maintained their mEOT-R. Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The number of participants with relapse was reported in treatment naive mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 960 | 518 | 427 | 128 | 11 | 4
percentage of participants
  24Wk PEOT, PEG-IFN alfa-2a (n=508,364,282,69,8,2) | 28.7 | 11.3 | 14.2 | 29.0 | 25.0 | 0
  24wk PEOT, PEG-IFN alfa-2b (n=91,93,57,7,2,0) | 20.9 | 7.5 | 10.5 | 28.6 | 15.0 | 0
Statistical Analysis 1: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 1.957, 95% CI 2-sided [1.383 to 2.770]
Statistical Analysis 2: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (< 140 vs >=180). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 3.337, 95% CI 2-sided [1.661 to 6.705]
Statistical Analysis 3: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (>=140 - < 180 vs >=180). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.3611, Regression, Logistic; Odds Ratio (OR) = 1.305, 95% CI 2-sided [0.737 to 2.312]
Statistical Analysis 4: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.943, 95% CI 2-sided [0.929 to 0.958]
Statistical Analysis 5: Comparison: Genotype 1 (G1); The statistical analysis is presented for cumulative ribavirin dose per 10000 mg, during the first 12 weeks. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 0.743, 95% CI 2-sided [0.615 to 0.897]
Statistical Analysis 6: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.864, 95% CI 2-sided [1.322 to 2.628]
Statistical Analysis 7: Comparison: Genotype 1 (G1); The statistical analysis is presented for mode of infection (other vs injection drug U). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0386, Regression, Logistic; Odds Ratio (OR) = 2.124, 95% CI 2-sided [1.040 to 4.338]
Statistical Analysis 8: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (< 140 vs >=180). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 3.398, 95% CI 2-sided [1.722 to 6.706]
Statistical Analysis 9: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (>=140 - < 180 vs >=180). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.2769, Regression, Logistic; Odds Ratio (OR) = 1.372, 95% CI 2-sided [0.776 to 2.428]
Statistical Analysis 10: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.945, 95% CI 2-sided [0.931 to 0.960]
Statistical Analysis 11: Comparison: Genotype 2 (G2); The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.163, 95% CI 2-sided [1.078 to 1.256]
Statistical Analysis 12: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.0213, Regression, Logistic; Odds Ratio (OR) = 1.788, 95% CI 2-sided [1.091 to 2.932]
Statistical Analysis 13: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 0.903, 95% CI 2-sided [0.856 to 0.953]
Statistical Analysis 14: Comparison: Genotype 2 (G2); The statistical analysis is presented for cumulative ribavirin dose per 10000 mg, first 12 weeks. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0306, Regression, Logistic; Odds Ratio (OR) = 0.723, 95% CI 2-sided [0.538 to 0.970]
Statistical Analysis 15: Comparison: Genotype 2 (G2); The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 1.145, 95% CI 2-sided [1.061 to 1.236]
Statistical Analysis 16: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 6]; Test type: Superiority or Other; p = 0.0122, Regression, Logistic; Odds Ratio (OR) = 1.907, 95% CI 2-sided [1.151 to 3.158]
Statistical Analysis 17: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 8]; Test type: Superiority or Other; p = 0.0956, Regression, Logistic; Odds Ratio (OR) = 2.175, 95% CI 2-sided [0.872 to 5.424]
Statistical Analysis 18: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 9]; Test type: Superiority or Other; p = 0.0846, Regression, Logistic; Odds Ratio (OR) = 0.267, 95% CI 2-sided [0.060 to 1.197]
Statistical Analysis 19: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 10]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.897, 95% CI 2-sided [0.852 to 0.945]
Statistical Analysis 20: Comparison: Genotype 3 (G3); The statistical analysis is presented for age per 10 years. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 1.996, 95% CI 2-sided [1.259 to 3.165]
Statistical Analysis 21: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 11]; Test type: Superiority or Other; p = 0.0095, Regression, Logistic; Odds Ratio (OR) = 1.150, 95% CI 2-sided [1.035 to 1.277]
Statistical Analysis 22: Comparison: Genotype 3 (G3); The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0031, Regression, Logistic; Odds Ratio (OR) = 0.155, 95% CI 2-sided [0.045 to 0.533]
Statistical Analysis 23: Comparison: Genotype 3 (G3); The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0645, Regression, Logistic; Odds Ratio (OR) = 0.364, 95% CI 2-sided [0.125 to 1.063]
Statistical Analysis 24: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 4]; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.895, 95% CI 2-sided [0.846 to 0.948]
Statistical Analysis 25: Comparison: Genotype 3 (G3); The statistical analysis is presented for age per 10 years. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 1.996, 95% CI 2-sided [1.259 to 3.165]
Statistical Analysis 26: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 15]; Test type: Superiority or Other; p = 0.0095, Regression, Logistic; Odds Ratio (OR) = 1.150, 95% CI 2-sided [1.035 to 1.277]
Statistical Analysis 27: Comparison: Genotype 3 (G3); The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0031, Regression, Logistic; Odds Ratio (OR) = 0.155, 95% CI 2-sided [0.045 to 0.533]
Statistical Analysis 28: Comparison: Genotype 3 (G3); The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0645, Regression, Logistic; Odds Ratio (OR) = 0.364, 95% CI 2-sided [0.125 to 1.063]
Statistical Analysis 29: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 10]; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.895, 95% CI 2-sided [0.846 to 0.948]
Statistical Analysis 30: Comparison: Genotype 1 (G1); The statistical analysis is presented for age per 10 years. The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0182, Regression, Logistic; Odds Ratio (OR) = 1.266, 95% CI 2-sided [1.041 to 1.541]
Statistical Analysis 31: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0092, Regression, Logistic; Odds Ratio (OR) = 1.590, 95% CI 2-sided [1.122 to 2.254]
Statistical Analysis 32: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (< 140 vs >=180). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 2.974, 95% CI 2-sided [1.488 to 5.942]
Statistical Analysis 33: Comparison: Genotype 1 (G1); The statistical analysis is presented for Platelets x 10**9/L at BL (>=140 - < 180 vs >=180). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.6524, Regression, Logistic; Odds Ratio (OR) = 1.142, 95% CI 2-sided [0.641 to 2.035]
Statistical Analysis 34: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (RVR vs No RVR/EVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.108, 95% CI 2-sided [0.037 to 0.311]
Statistical Analysis 35: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (cEVR vs No RVR/EVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0429, Regression, Logistic; Odds Ratio (OR) = 0.389, 95% CI 2-sided [0.156 to 0.970]
Statistical Analysis 36: Comparison: Genotype 1 (G1); The statistical analysis is presented for on-treatment response (pEVR vs No RVR/EVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.5490, Regression, Logistic; Odds Ratio (OR) = 1.330, 95% CI 2-sided [0.523 to 3.380]
Statistical Analysis 37: Comparison: Genotype 2 (G2); The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for relapse was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 1.136, 95% CI 2-sided [1.054 to 1.224]
Statistical Analysis 38: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 31]; Test type: Superiority or Other; p = 0.0140, Regression, Logistic; Odds Ratio (OR) = 1.855, 95% CI 2-sided [1.133 to 3.037]
Statistical Analysis 39: Comparison: Genotype 2 (G2); The statistical analysis is presented for on-treatment response (RVR vs No RVR/EVR). The logistic regression analysis for relapse was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0575, Regression, Logistic; Odds Ratio (OR) = 0.126, 95% CI 2-sided [0.015 to 1.068]
Statistical Analysis 40: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 35]; Test type: Superiority or Other; p = 0.7128, Regression, Logistic; Odds Ratio (OR) = 0.660, 95% CI 2-sided [0.072 to 6.025]
Statistical Analysis 41: Comparison: Genotype 2 (G2); [analysis description as in outcome 21, analysis 36]; Test type: Superiority or Other; p = 0.5960, Regression, Logistic; Odds Ratio (OR) = 0.505, 95% CI 2-sided [0.040 to 6.318]
Statistical Analysis 42: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 30]; Test type: Superiority or Other; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 2.051, 95% CI 2-sided [1.270 to 3.311]
Statistical Analysis 43: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 37]; Test type: Superiority or Other; p = 0.0452, Regression, Logistic; Odds Ratio (OR) = 1.113, 95% CI 2-sided [1.002 to 1.236]
Statistical Analysis 44: Comparison: Genotype 3 (G3); The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for relapse was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0040, Regression, Logistic; Odds Ratio (OR) = 0.154, 95% CI 2-sided [0.043 to 0.551]
Statistical Analysis 45: Comparison: Genotype 3 (G3); The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for relapse was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0833, Regression, Logistic; Odds Ratio (OR) = 0.393, 95% CI 2-sided [0.137 to 1.131]
Statistical Analysis 46: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 39]; Test type: Superiority or Other; p = 0.1439, Regression, Logistic; Odds Ratio (OR) = 0.141, 95% CI 2-sided [0.010 to 1.951]
Statistical Analysis 47: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 35]; Test type: Superiority or Other; p = 0.4457, Regression, Logistic; Odds Ratio (OR) = 0.350, 95% CI 2-sided [0.024 to 5.194]
Statistical Analysis 48: Comparison: Genotype 3 (G3); [analysis description as in outcome 21, analysis 36]; Test type: Superiority or Other; p = 0.6258, Regression, Logistic; Odds Ratio (OR) = 2.142, 95% CI 2-sided [0.100 to 45.801]

22. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Per Protocol Population at 24 Weeks After End of Treatment
Description: as for outcome 20
Time Frame: At 24 weeks after EOT
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Number analyzed (Participants) | 862 | 448 | 367 | 116 | 9 | 4
percentage of participants
  24Wk PEOT, PEG-IFN alfa-2a (n=468,323,240,60,6,2) | 28.4 | 11.5 | 13.8 | 31.7 | 33.3 | 0
  24wk PEOT, PEG-IFN alfa-2b (n=79,77,53,7,2,0) | 21.5 | 7.8 | 11.3 | 28.6 | 50.0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks after EOT. The EOT is 12, 24, 48 or 72 weeks after initiation of treatment.
Description: Documentation of adverse events or serious adverse events was not within scope of this study. Serious Adverse Drug Reactions (SADRs) were reported through spontaneous reporting system for marketed drugs. In most SADRs, the study number was missing on form; thus it could not be assigned to study and hence no data was available for reporting.
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Unknown Genotype (UNK)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.